CLINICAL TRIAL: NCT05666622
Title: Can Delta Neutrophil Index Values Predict the Success of Periodontal Treatment in Patients With Periodontitis?
Brief Title: DNI Values After Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Eda Cetin Ozdemir, assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/18-05
Record Dates: First submitted 2022-12-09; First posted 2022-12-28 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis; Periodontal Inflammation; Inflammatory Response
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kahramanmaraş Sütçü İmam University (Other): Only routine non-surgical periodontal treatment was applied to the patients.
  Interventions: Other: Only routine non-surgical periodontal treatment was applied to the patients.

INTERVENTIONS:
Other: Only routine non-surgical periodontal treatment was applied to the patients. — The study included 70 systemically healthy individuals, as a test group of 35 patients with Stage 3, Grade A periodontitis and a control group of 35 individuals with no periodontal disease. Blood samples were taken for the examination of DNI, white blood cells (WBC), immature granulocytes (IG), procalcitonin, C-reactive protein (CRP), lymphocyte count and neutrophil count. For the patients with periodontitis, blood sample assays were repeated 3 months after non-surgical periodontal treatment

SUMMARY:
The study included 70 systemically healthy individuals, as a test group of 35 patients with Stage 3, Grade A periodontitis and a control group of 35 individuals with no periodontal disease. Blood samples were taken for the examination of DNI, white blood cells (WBC), immature granulocytes (IG), procalcitonin, C-reactive protein (CRP), lymphocyte count and neutrophil count. For the patients with periodontitis, blood sample assays were repeated 3 months after NSPT.

DETAILED DESCRIPTION:
The role of the Delta Neutrophil Index (DNI) in the pathogenesis and follow-up of periodontal disease has not been comprehensively documented. The study included 70 systemically healthy individuals, as a test group of 35 patients with Stage 3, Grade A periodontitis and a control group of 35 individuals with no periodontal disease. Blood samples were taken for the examination of DNI, white blood cells (WBC), immature granulocytes (IG), procalcitonin, C-reactive protein (CRP), lymphocyte count and neutrophil count. For the patients with periodontitis, blood sample assays were repeated 3 months after NSPT.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis
* Patients have more than 20 teeth in the mouth
* Minimum age 18
* Maximum age 65

Exclusion Criteria:

* Patients with any systemic disease
* Active smokers
* Pregnant or breastfeeding
* Patients have used any antibiotic or anti-inflammatory drug in the last 6 months
* Patients have received any periodontal treatment in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in Delta Neutrophil Index values of periodontal treatment in patients with periodontitis. | 12 weeks
  We expect a decrease in the Delta Neutrophil Index values after non-surgical periodontal treatment.

SECONDARY OUTCOMES:
Neutrophil-lymphocyte ratio (NLR) values after non-surgical periodontal treatment. | 12 weeks
  We expect a decrease in the neutrophil-lymphocyte ratio (NLR) values after non-surgical periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Çetin Özdemir, Dr., Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts FA, Darveau RP. Microbial protection and virulence in periodontal tissue as a function of polymicrobial communities: symbiosis and dysbiosis. Periodontol 2000. 2015 Oct;69(1):18-27. doi: 10.1111/prd.12087. PMID 26252399
- [Background] Hajishengallis G. Periodontitis: from microbial immune subversion to systemic inflammation. Nat Rev Immunol. 2015 Jan;15(1):30-44. doi: 10.1038/nri3785. PMID 25534621
- [Background] Hajishengallis G, Chavakis T. Local and systemic mechanisms linking periodontal disease and inflammatory comorbidities. Nat Rev Immunol. 2021 Jul;21(7):426-440. doi: 10.1038/s41577-020-00488-6. Epub 2021 Jan 28. PMID 33510490
- [Background] Acharya AB, Shetty IP, Jain S, Padakannaya I, Acharya S, Shettar L, Thakur S. Neutrophil-to-lymphocyte ratio and platelet-to-lymphocyte ratio in chronic periodontitis before and after nonsurgical therapy. J Indian Soc Periodontol. 2019 Sep-Oct;23(5):419-423. doi: 10.4103/jisp.jisp_622_18. PMID 31543614
- [Background] Valiyaveetil Karattil L, Joseph RS, Ambooken M, Mathew JJ. Evaluation of serum concentrations of hs-CRP and Hb in varying severities of chronic periodontitis. Biomarkers. 2022 May;27(3):258-263. doi: 10.1080/1354750X.2022.2032349. Epub 2022 Feb 2. PMID 35060836
- [Background] Yoon NB, Son C, Um SJ. Role of the neutrophil-lymphocyte count ratio in the differential diagnosis between pulmonary tuberculosis and bacterial community-acquired pneumonia. Ann Lab Med. 2013 Mar;33(2):105-10. doi: 10.3343/alm.2013.33.2.105. Epub 2013 Feb 21. PMID 23482854
- [Derived] Ozdemir EC, Bozkurt E, Yazar FM, Bozan MB. Can delta neutrophil index values predict the success of periodontal treatment in patients with periodontitis? Clin Oral Investig. 2024 Jan 9;28(1):82. doi: 10.1007/s00784-023-05478-1. PMID 38195732